CLINICAL TRIAL: NCT05348018
Title: Implementation of Game-based Training in Oral Rehabilitation of Edentulous Patients in Undergraduate Dental Course
Brief Title: Serious Games for Training in Oral Rehabilitation
Acronym: Playdent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Rothschild (Other)
Responsible Party: Principal Investigator, Dr Braud Adeline, Professor, Hôpital Rothschild
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PlY01
Record Dates: First submitted 2022-04-19; First posted 2022-04-27 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Health Knowledge, Attitudes, Practice
Keywords: health education
MeSH Terms: conditions — Behavior; Health Education

STUDY DESIGN:
Intervention Model Description: Participants were allocated either to a "test" group which accessed Serious games during a four-week test period in addition to conventional lectures or to a "control" group which benefited solely from conventional lectures
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "test" group (Experimental): "test" group which accessed SGs during a four-week test period in addition to conventional lectures
  Interventions: Device: Playing Serious Games during a four-week test period in addition to conventional lectures
- "control" group (No Intervention): "control" group which benefited solely from conventional lectures

INTERVENTIONS:
Device: Playing Serious Games during a four-week test period in addition to conventional lectures — Playing SGs during a four-week test period in addition to conventional lectures in oral rehabilitation
  Arms: "test" group

SUMMARY:
Coronavirus disease-19 (COVID-19) dramatically changed the learning conditions of dental students, with restricted access to training sessions and clinical practice. The "Playdent" project proposed the integration of serious games (SGs) in the third-year curriculum, based on tailor-made scenarios questioning the first dental visit of edentulous patients, and examined whether training with the games would advance students' learning outcomes.

DETAILED DESCRIPTION:
Three Serious games proposed in addition to conventional lectures and practical exercises in oral rehabilitation of edentulous patients were supposed to improve knowledge and skills of undergraduates. However, in order to assess the influence of SGs on students' learning outcomes and subsequent satisfaction, a single-blind controlled protocol was designed. The null hypothesis was that SGs had no impact on the learning outcomes of undergraduate students.

ELIGIBILITY:
Inclusion Criteria:

* adult students (aged at least 18)
* enrolled in the third-year at the faculty of dental surgery of the University of Paris,
* agreeing to participate in the study

Exclusion Criteria:

* Third-year students who had repeated their courses

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
performance | One month
  Students' performance for managing a dental visit of edentulous patients were assessed by measuring score to a test developed by the teaching team. Scores were calculated ranging from 0 (no correct answer) to 15 (100% correct answers).

SECONDARY OUTCOMES:
students' satisfaction | one month
  a questionnaire was drawn up for the students in the form of an self-administered questionnaire, which included questions pertaining to their satisfaction ranging from 0 (=very unsatisfactory) to 10 (=very satisfactory).

CONTACTS AND LOCATIONS:
Overall Officials: Adeline Braud, PhD, Principal Investigator — Unievrsité de Paris
Locations (1):
- Université de Paris, Paris, Parisl, France

IPD SHARING:
Plan to Share IPD: No